CLINICAL TRIAL: NCT07042100
Title: A Phase 1, Multicentre, Open-label, Multiple-dose Study to Determine Safety, Tolerability, and Preliminary Efficacy of SBO-154 in Subjects With Advanced Solid Tumors
Brief Title: A Study to Test the Safety and Tolerability of SBO-154 in Patients With Advanced Solid Tumors.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SBO-154-25-01
Record Dates: First submitted 2025-05-28; First posted 2025-06-27 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SBO-154 (Experimental)
  Interventions: Biological: Dose level (DL)1; Biological: DL2; Biological: DL3; Biological: DL4; Biological: DL5

INTERVENTIONS:
Biological: Dose level (DL)1 — Administered IV every 3 weeks
Biological: DL2 — Administered IV every 3 weeks
Biological: DL3 — Administered IV every 3 weeks
Biological: DL4 — Administered IV every 3 weeks
Biological: DL5 — Administered IV every 3 weeks

SUMMARY:
This is a Phase 1 study of SBO-154 in patients with advanced cancers who are unable to tolerate or have not previously responded to standard therapy available in the country. The study involves multiple doses and takes place at several centers.

DETAILED DESCRIPTION:
This study has two parts. In Part 1, the goal to evaluate the safety and tolerability along with the highest dose that can be tolerated, or the dose(s) which can be chosen for further evaluation. In Part 2, the focus is on evaluating the safety of SBO-154 in specific types of advanced cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written and dated informed consent (or legally acceptable representative/ impartial witness when applicable) and is available for the entire study.
2. Willing and able to comply with the scheduled visits, treatment plan, laboratory testing, study procedures, and restrictions (in the Investigator's opinion), and be accessible for follow-up.
3. Has locally recurrent or metastatic disease (except sarcomas) which has relapsed or progressed following local standard treatment, or for which no standard treatment is available.
4. Has a life expectancy of ≥3 months.

Exclusion Criteria:

1. Any major surgery, as determined by the Investigator, within 4 weeks of SBO-154 administration.
2. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination.
3. Known or suspected history of significant drug abuse as judged by the Investigator.
4. Has an uncontrolled infection requiring intravenous (IV) antibiotics, antivirals, or antifungals.
5. Known or suspected history of excessive intake of alcohol in the 12 months prior to study entry.
6. Positive exclusion tests: urine pregnancy tests (if applicable), serology tests positive for HIV, HCV, HBsAg (unless they are considered subjects with resolved Hepatitis B and C infection).
7. History of any relevant allergy/ hypersensitivity including known immediate or delayed hypersensitivity reaction or idiosyncrasy to biological agents or drug chemically related to SBO-154 or its excipients.
8. Received an investigational agent within 30 days or 5 half-lives- whichever is shorter prior to SBO-154 administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities | Twenty-one days from the initiation of the first dose of SBO-154 (3 weeks)
  Applicable to Part 1 only
Incidence of treatment-related serious adverse events | Throughout the study: from the start of study drug to 30 days post the last dose of study drug.
Incidence of treatment-related adverse events | Throughout the study: from the start of study drug to 30 days post the last dose of study drug.

SECONDARY OUTCOMES:
To evaluate the overall response rate (i.e., the percentage of participants who achieved a best response of Complete Response (CR) or Partial Response (PR), per RECIST v1.1) | Time Frame: Assessed every 6 weeks from the date of first study drug administration until the date of first documented disease progression, or death, whatever comes first; assessed for an average of 12 months.
To evaluate the duration of response (i.e., the time from the initial response (CR or PR) to the time of progression of disease (PD) or death, per RECIST v1.1) | Time Frame: Assessed every 6 weeks from the date of first study drug administration until the date of first documented disease progression, or death, whatever comes first; assessed for an average of 12 months.
To evaluate the disease control rate (i.e., the percentage of participants who achieved a best response of CR, PR, or remained stable disease (SD), per RECIST v1.1) | Time Frame: Assessed every 6 weeks from the date of first study drug administration until the date of first documented disease progression, or death, whatever comes first; assessed for an average of 12 months.
To evaluate the time to response (i.e., the time from treatment start to the time-point where a best response of CR or PR was achieved, per RECIST v1.1) | Time Frame: Assessed every 6 weeks from the date of first study drug administration until the date of first documented disease progression, or death, whatever comes first; assessed for an average of 12 months.
To evaluate the progression-free survival (i.e., the time from treatment start to the time of PD or death, per RECIST v1.1) | Time Frame: Assessed every 6 weeks from the date of first study drug administration until the date of first documented disease progression, or death, whatever comes first; assessed for an average of 12 months.
Incidences of anti-drug antibodies (ADA) | Survival Follow-up: Upto 1 yr
Incidences of titer antibodies | Survival Follow-up: Upto 1 yr
Incidences of neutralizing antibodies | Survival Follow-up: Upto 1 yr

CONTACTS AND LOCATIONS:
Locations (11):
- United States (5):
  - Honorhealth Research Institute, Scottsdale, Arizona
  - Sarcoma Oncology Research Center, Santa Monica, California
  - Yale University - Yale Cancer Center, New Haven, Connecticut
  - Hope And Healing Cancer Services, Llc, Hinsdale, Illinois
  - MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Scientia Clinical Research, Randwick, New South Wales
  - Sunshine Coast University Private Hospital, Birtinya, Queensland
  - Cancer Research South Australia, Adelaide, South Australia
- India (3):
  - Tata Memorial hospital, Mumbai, Maharashtra
  - Noble Hospital Pvt. Ltd., Pune, Maharashtra
  - All India Institute for Medical Sciences, Delhi, New Delhi

IPD SHARING:
Plan to Share IPD: No